CLINICAL TRIAL: NCT04710290
Title: A Cohort Study to Evaluate the Efficacy of Beta-Glucan or Beta-Glucan Compound (Combined With Glutamine and Immunoglobulin) Supplement in Patients With Metastatic Cancers Undergoing Chemotherapy
Brief Title: A Cohort Study of Beta-Glucan or Beta-Glucan Compound in Metastatic Cancers
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: E-DA Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EMRP50106N
Record Dates: First submitted 2020-01-05; First posted 2021-01-14 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Metastatic Cancer; Chemotherapy
Keywords: beta-glucan; metastatic cancer; chemotherapy
MeSH Terms: conditions — Neoplasm Metastasis | interventions — beta-Glucans; Glutamine; Starch

STUDY DESIGN:
Intervention Model Description: beta-glucan group; beta-glucan + glutamin; placebo
Who Masked: Participant
Masking Description: this trial is single-blind clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Solid beverage powder (Experimental): Whey portein solid beverage powder use 1 pack for every 10 kg of body weight. A total of 6 pack under 60 kg a day, an extra 1pack for each additional 10 kg over 60 kg.Use from the 7th day of the 2nd course of treatment for 5 months.
  Interventions: Dietary Supplement: Beta-Glucan; Dietary Supplement: Glutamine; Dietary Supplement: Immunoglobuin
- Capsule (Experimental): Capsules use 1 cap for every 10 kg of body weight.A total of 6 cap under 60 kg a day, an extra 1cap for each additional 10 kg over 60 kg. Use from the 7th day of the 2nd course of treatment for 5 months.
  Interventions: Dietary Supplement: Beta-Glucan
- Placebo (Placebo Comparator): placebo use 1 powder for every 10 kg of body weight. A total of 6 pack under 60 kg a day, an extra 1pack for each additional 10 kg over 60 kg.Use from the 7th day of the 2nd course of treatment for 5 months.
  Interventions: Dietary Supplement: Corn starch

INTERVENTIONS:
Dietary Supplement: Beta-Glucan — Solid beverage powders, capsules and placebo were randomly assigned. The main components of the solid beverage powder are beta-glucan combined with glutamine and immunoglobuin.and the main component of the capsule is beta-glucan . The main ingredient of placebo is corn starch.
  Arms: Capsule; Solid beverage powder
Dietary Supplement: Glutamine — Solid beverage powders, capsules and placebo were randomly assigned. The main components of the solid beverage powder are beta-glucan combined with glutamine and immunoglobuin.and the main component of the capsule is beta-glucan . The main ingredient of placebo is corn starch.
  Arms: Solid beverage powder
Dietary Supplement: Immunoglobuin — Solid beverage powders, capsules and placebo were randomly assigned. The main components of the solid beverage powder are beta-glucan combined with glutamine and immunoglobuin.and the main component of the capsule is beta-glucan . The main ingredient of placebo is corn starch.
  Arms: Solid beverage powder
Dietary Supplement: Corn starch — Solid beverage powders, capsules and placebo were randomly assigned. The main components of the solid beverage powder are beta-glucan combined with glutamine and immunoglobuin.and the main component of the capsule is beta-glucan . The main ingredient of placebo is corn starch.
  Arms: Placebo

SUMMARY:
Immunity of cancer patients is an important issue. According to cancer immunity, it can be divided into three phases: clearance phase, equilibrium phase, and escape phase (cancer cells can avoid the recognition of immune cells). Βeta-glucans is extracted from yeast, it can increase immune function and drive of hematopoietic stem cells in animals and clinical trials. Glutamine can increase the repair of oral and intestinal mucosa of patients receiving chemical and radiation therapy and can increase the lymphocytes of patients. Colostrum contains IgA, IgG, IgM, etc., known to protect the baby Cancer patients who are infected with intestinal bacteria and undergo systemic chemotherapy are less immune than normal adults.

Investigators will compare β-glucan, glutamine, and colostrum immunoglobulin powder with β-glucan and control group, each group has 30 people, and observe the side effects and blood of patients under standard chemotherapy. The performance of the immune system, such as helpers and cytotoxic T cells and NK cells, and to observe the differences in treatment interruption or delay rates and treatment rates.

DETAILED DESCRIPTION:
Experiment theme / background:

Cancer immune surveillance is considered to be an important host protection process to inhibit carcinogenesis and to maintain cellular homeostasis. In the interaction of host and tumor cells, three essential phases have been proposed: elimination, equilibrium, and escape.

In the elimination stage, a small portion of cancer cells can be eliminated by immune reactions. Direct cancer and innate immune system interaction including natural killer cells (NK), dendritic cells (DC), macrophages, polymorphonuclear leukocytes (PM including neutrophils, eosinophils, and basophils), mast cells and cytotoxic T lymphocytes, directly target cancer cells. NK cells, DC, PMN, mast cells, and macrophages are first-line effectors to damaged cells and cancer cells. NK-T cells and γδ T cells play roles as both innate and adaptive components, through close interactions with cells of the adaptive immune system, such as CD4+ and CD8+ T lymphocytes with cytotoxic effects and memory. In addition to direct cancer/innate immune system interactions, a large number of molecules released due to cancer cell death, may function as damage-associated molecular patterns (DAMP) and interact with innate immune cells. Those cancer-derived DAMP include both intracellular molecules and extracellular matrix (ECM) molecules released from apoptotic and necrotic tumor cells.

However, cancer cells show immune tolerance and go in to escape stage. Currently, programmed death-1 (PD-1) in T cells and programmed death ligands 1 and 2 in cancer cells overexpression was proved as one of the mechanisms of immune tolerance of cancer cells. The cytotoxic T-lymphocyte-associated antigen -4 (CTLA-4) is another negative regulator of immune reaction in cancer patients. Immune therapy including anti-PD1, anti-PD-L1, anti-CTLA4 medicines, developed and showed clinical benefit in many cancer types, including melanoma, renal cell carcinoma, head and neck cancer, non-small cell lung cancer, etc. It shows us that if investigators can break immune tolerance in cancer patients, cancer can be controlled.

Beta-glucan (long polymer ([1,6] B-d-glucopyranosoyl-[1,3] Bd-glucopyranose, PGG) is isolated from Baker's yeast (Saccharomyces cerevisiae).8 Preparation of purified yeast beta-glucan sphere is commercially available in the form of whole glucan particles (Wellmune, WGPs) as a food supplement. Further efforts resulted in the development of a water-soluble, pharmaceutical-grade yeast beta-glucan whose biological effects have been extensively studied in vivo. Beta-glucan particle is consumed by macrophages after being transported from the lumen of the small intestine through Peyer's patches. The macrophage degrades the beta-glucan (a pro-drug) to its bioactive fractions.

Two major functions of beta-glucan are immune stimulation and hematopoietic stem cell mobilization. A substantial number of studies have indicated that beta-glucan functions to increase the host immune response to infection and cancer Small molecular weight WGPs exert their function through neutrophils by priming complement receptor 3 (CR3) to kill iC3b-opsonized microorganism or tumor cells. The complement (C) system is a major component of innate immunity and plays a critical role in host defense, but also enhances adaptive immunity through the regulation of both T- and B-cell responses. Furthermore, GPS elicit mouse dendritic cells to release a significantly higher amount of IL-12 but a lower amount of IL-6 and TNF, as a potent promoter of Th1 adaptive responses. Cellular immunity against tumor cells chiefly is dependent on Th1 immune responses.

Early studies of WGPs demonstrated a rapid hematopoietic recovery following bone marrow injury from irradiation and chemotherapeutic agents. Stem-cell mobilizing effects of WGP and the combination of WGP with G-CSF have been studied. A single dose of WGP beta-glucan was found to mobilize hematopoietic progenitor cells (HPCs) to the peripheral blood. Moreover, an additive effect was seen when WGP beta-glucan was used in conjunction with G-CSF. This mobilization ability requires the activity of matrix metalloproteinase. Because hematopoietic stem cell mobilization is enhanced by beta-glucan, WGP is able to shorten the leucopenia period of patients after chemotherapy. Patients undertaking treatment with WGP should have a better quality of life (QoL) because higher immunity and leukocyte level are essential to prevent infection after chemotherapy.

A significant amount of pre-clinical and clinical data is available supporting the efficacy of this product. A clinical study of advanced colorectal cancer treated with FORFIRI plus Cetuximab compared to FORFIRI/Cetuximab/beta-glucan has been reported in the ASCO annual meeting.23 Median progression-free survival increased 38% to 22 weeks with the beta-glucan combination, compared with 16 weeks for the standard of care. The overall response rate (complete response + partial response) was 30% with beta-glucan combination, compared to 16% for the standard of care.

Glutamine is an abundant and versatile nutrient that participates in energy formation, redox homeostasis, macromolecular synthesis, and signaling in cancer cells. Glutamine levels in plasma and skeletal muscle were decreased in tumor-bearing rats, although glutamine production and the conversion of arginine to glutamine were increased. Glutamine supplement reduced whole-body protein breakdown rate during chemotherapy in tumor-bearing rats and increase fat-free mass in cancer-related cachexia patients. It also enhanced lymphocyte mitogenic function and reduced permeability of the gut during radiochemotherapy in esophageal cancer patients. However, the role of glutamine in cancer growth is equivocal. In some cancer cells, excess glutamine is exported in exchange for leucine and other essential amino acids. This exchange facilitates activation of the serine/threonine kinase mTOR, a major positive regulator of cell growth. An opposite study showed that glutathione (GSH) increases under glutamine supplementation that can resist chemotherapy and radiotherapy in normal cells. In cancer tissue, glutamine supplementation appears to decrease intratumoral GSH stores, which may cause sensitivity to treatment.

Test purposes:

Investigators need to evaluate the efficacy of bone marrow function recovery after chemotherapy, analyze the type of immune cells, and measure the number of immune cells, including CD4 + T cells, CD8 + T cells, NK-T cells, etc., which can help innate immune response, cancer response. In addition, Investigators want to assess whether simultaneous treatments can help treat response and quality of life.

Experiment method:

Study nutritional supplements have been used since the 7th day of Week 2 and lasted to 2 months after completing 6 cycles of systemization, using one pack or one nutrient for every 10 kg of body weight Tracking or rehabilitation plan: The case is closed for one year, and the case is tracked one year after the case is closed. On the seventh day of the second course, on the twenty-first day, on the seventh day of the fourth course, on the twenty-second day of the sixth course, and two months after the end of the treatment, 10 c.c. of blood were taken for the leukocyte surface antigen test, and in the second course The seventh day, the fourth course of treatment, the seventh day, the sixth course of the 22nd day.

Main efficacy or evaluation index: When the subjects joined the trial, the clinician's treatment needs a complete examination, including the detection of hepatitis B surface antigen and hepatitis C antibody, on the seventh day of the second course, the twenty-first day, and the seventh day of the fourth course On the 22nd day of the 6th course of treatment, and taking 10cc of blood for two weeks to complete the leukocyte surface antigen test two months after the treatment, And two months after the end of treatment and assisted in the assessment of the quality of life scale (with EORTC QLQ-C30 and QLQ-CX24 Taiwan Chinese version)

Primary endpoint:

* 1. Assess the white blood cell status of the three groups of patients before, after and two months after the end of chemotherapy,

Including the distribution and performance of T cells, B cells, and NK cells.

* 2. Improvement of patients' quality of life.

Secondary endpoint

* 1. The smoothness of patient treatment, such as whether to receive treatment as scheduled and whether there is an infection.
* 2. Overall survival and no-deterioration survival.

Statistical methods:

* 1. Evaluation with Quality of Life Scale (with EORTC QLQ-C30 and QLQ-CX24 Taiwanese Chinese version)
* 2. Use regression analysis to analyze the white blood cells of the three groups of patients before, after and two months after the end of chemotherapy. Conditions, including the distribution and performance of T cells, B cells and NK cells.
* 3. Kaplan Meunier survival curve analysis of overall survival and non-deterioration survival.

Possible harm criteria:

According to the results of current trials and clinical use of this nutritional supplement, no obvious side effects have been found, but patients with lactose intolerance may experience mild diarrhea, which can be reduced or discontinued; very few people may produce Allergic reactions or glutamic acid, if there have been allergic reactions such as rash, immediately withdraw from the test.

Processing method:

When the subject has any discomfort, please tell the subject's trial host doctor, the doctor will try his best to give the subject the best treatment and care. If the subject has any emergency or other unusual physical condition, which cannot be effectively controlled with existing drugs, please contact the subject's physician immediately. When the subject encounters serious side effects or complications on a regular holiday, please immediately send it to the emergency room of the subject's hospital and inform the emergency physician of the content of the human trial he participated in.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic cancer receiving systemic chemotherapy
* ECOG=0,1
* Age ≥20 years
* Chemotherapy drugs include platinum drugs (cisplatin, carboplatin, oxaliplatin), irinotecan / topotecan, paclitaxel (docetaxel), fluorouracil (5-FU), and alkylating drugs (such as cyclophosphamide)

Exclusion Criteria:

* Early cancer patients.
* Patients receiving systemic chemotherapy or large-area radiation therapy 6 months before chemotherapy.
* The patient had a history of allergies to β-glucan or glutamine.
* Patients with liver dysfunction not associated with cancer. (GOT> 2 × ULN; GPT> 2 × ULN)
* Patients with abnormal renal function (creatinine over 2 mg / dl)
* Age <20 years

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-01-04 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
the change of total white blood cells, neutrophils, and lymphocytes at day 14 of 2nd cycle, from day 7 of 2nd cycle of chemotherapy | 7days
  the units of white blood cells, neutrophils, and lymphocytes are /ul.
the change of total white blood cells, neutrophils, and lymphocytes at day 1 of 3rd cycle, from day 14 of 2nd cycle of chemotherapy | 14-21 days
  the units of white blood cells, neutrophils, and lymphocytes are /ul
the change of total white blood cells, neutrophils, and lymphocytes at day 7 of 3rd cycle, from day 1 of 3rd cycle of chemotherapy | 7 days
  the units of white blood cells, neutrophils, and lymphocytes are /ul.
the change of total white blood cells, neutrophils, and lymphocytes at day 7 of 4th cycle, from day 7 of 3rd cycle of chemotherapy | 21-28 days
  the units of white blood cells, neutrophils, and lymphocytes are /ul.
the change of total white blood cells, neutrophils, and lymphocytes at day 1 of 5th cycle, from day 7 of 4th cycle of chemotherapy | 14-21 days
  the units of white blood cells, neutrophils, and lymphocytes are /ul.
the change of total white blood cells, neutrophils, and lymphocytes at day 7 of 5th cycle, from day 1 of 5th cycle of chemotherapy | 7 days
  the units of white blood cells, neutrophils, and lymphocytes are /ul.
the change of total white blood cells, neutrophils, and lymphocytes at day 1 of 6th cycle, from day 7 of 5th cycle of chemotherapy | 14-21 days
  the units of white blood cells, neutrophils, and lymphocytes are /ul.
the change of total white blood cells, neutrophils, and lymphocytes at day 7 of 6th cycle, from day 1 of 6th cycle of chemotherapy | 7 days
  the units of white blood cells, neutrophils, and lymphocytes are /ul.
the change of total white blood cells, neutrophils, and lymphocytes at day 22 of 6th cycle, from day 7 of 6th cycle of chemotherapy | 15 days
  the units of white blood cells, neutrophils, and lymphocytes are /ul.
the change of total white blood cells, neutrophils, and lymphocytes at 2nd month after chemotherapy, from day 22 of 6th cycle of chemotherapy | 63 days
  the units of white blood cells, neutrophils, and lymphocytes are /ul.
change of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30) and EORTC-quality-of-life questionnaire cervical cancer module (EORTC-QLQ-CX24 [Taiwan version]) score at C4D7 from C2D7 | 6-8 weeks
  total 54 questions. 1-4 points for each EORTC QLQ-C30 and EORTC QLQ-CX24 (Taiwan version) are continue question list, that contain total 54 questions.
  The questionnaire is divided into two parts.One is that the higher the score, the more obvious the uncomfortable symptoms.One is that the higher the score, the better the state, for example:1. The overall health score of the self-assessment in this week is 7 points, 1 point means very poor and 7 points means excellent.2. Self-assess the overall quality of life during the week. 1 point means very poor and 7 points means excellent.
change of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30) and EORTC-quality-of-life questionnaire cervical cancer module (EORTC-QLQ-CX24 [Taiwan version]) score at C6D22 from C4D7 | 8-10 weeks
  total 54 questions. 1-4 points for each EORTC QLQ-C30 and EORTC QLQ-CX24 (Taiwan version) are continue question list, that contain total 54 questions The questionnaire is divided into two parts.One is that the higher the score, the more obvious the uncomfortable symptoms.One is that the higher the score, the better the state, for example:1. The overall health score of the self-assessment in this week is 7 points, 1 point means very poor and 7 points means excellent.2. Self-assess the overall quality of life during the week. 1 point means very poor and 7 points means excellent.
change of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30) and EORTC-quality-of-life questionnaire cervical cancer module (EORTC-QLQ-CX24 [Taiwan version]) score at 2 month from C6D22 | 9 -10 weeks
  total 54 questions. 1-4 points for each EORTC QLQ-C30 and EORTC QLQ-CX24 (Taiwan version) are continue question list, that contain total 54 questions The questionnaire is divided into two parts.One is that the higher the score, the more obvious the uncomfortable symptoms.One is that the higher the score, the better the state, for example:1. The overall health score of the self-assessment in this week is 7 points, 1 point means very poor and 7 points means excellent.2. Self-assess the overall quality of life during the week. 1 point means very poor and 7 points means excellent.
the change of lymphocyte surface markers percentage at day 7 of 2nd chemotherapy, from baseline. | 4-5 weeks
  the lymphocytes surface markers including:CD3, CD4, CD8, CD20, CD28, CD279, CD16, CD56, CD158a/h, CD158b, CD158e, CD158f, CD158i
the change of lymphocyte surface markers percentage at day 14 of 2nd chemotherapy, from day 7 of 2nd chemotherapy | 7 days
  the lymphocytes surface markers including:CD3, CD4, CD8, CD20, CD28, CD279, CD16, CD56, CD158a/h, CD158b, CD158e, CD158f, CD158i
the change of lymphocyte surface markers percentage at day 7 of 4th cycle of chemotherapy, from day 14 of 2nd chemotherapy | 5-7 weeks
  the lymphocytes surface markers including:CD3, CD4, CD8, CD20, CD28, CD279, CD16, CD56, CD158a/h, CD158b, CD158e, CD158f, CD158i
the change of lymphocyte surface markers percentage at day 22 of 6th cycle of chemotherapy, from day 7 of 4th cycle of chemotherapy | 8-10 weeks
  the lymphocytes surface markers including:CD3, CD4, CD8, CD20, CD28, CD279, CD16, CD56, CD158a/h, CD158b, CD158e, CD158f, CD158i
the change of lymphocyte surface markers percentage at 2 month after 6th cycle of chemotherapy, from day 22 of 6th cycle of chemotherapy | 5 weeks
  the lymphocytes surface markers including:CD3, CD4, CD8, CD20, CD28, CD279, CD16, CD56, CD158a/h, CD158b, CD158e, CD158f, CD158i

SECONDARY OUTCOMES:
analysis overall survival | 2 years
  we will follow up overall survival of patients in 3 groups until 2 years after the last patient enroll.

CONTACTS AND LOCATIONS:
Locations (1):
- E-DA hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No